CLINICAL TRIAL: NCT00002166
Title: An Open-Label, Non-Randomized Trial to Evaluate the Tolerability and Safety of Viramune (Nevirapine) in Adult and Pediatric Patients With Progressive HIV Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 200D; 1100.859
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-08

CONDITIONS: HIV Infections
Keywords: Nevirapine; Reverse Transcriptase Inhibitors; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine

INTERVENTIONS:
Drug: Nevirapine

SUMMARY:
To provide access to Viramune and to evaluate the tolerance and safety of Viramune in patients with progressive, symptomatic HIV disease who failed or are intolerant to currently approved treatment for HIV-1 infection and who are unable to participate in another Viramune controlled clinical trial and have a compelling need for anti-HIV treatment.

DETAILED DESCRIPTION:
Eligible adult patients (>= 13 years of age) will receive treatment with Viramune once daily for 2 weeks and then twice daily. Eligible pediatric patients (< 13 years of age) will receive a lower dose of Viramune once daily for 2 weeks and then twice daily. All patients will receive Viramune with or without concomitant antiretroviral therapy. Patients will be evaluated at weeks 2, 4, 8, 16, 24, 32 and every 8 weeks thereafter.

PER AMENDMENT 01/31/97: Enrollment closed to adult patients. As of 1/31/97 only enrolling pediatric patients.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Patients > 18 months of age with history of positive serology for HIV-1 infection or patients <= 18 months of age with history of positive viral culture, detectable p24 antigen, or positive peripheral blood mononuclear cell macro culture.
* Patients >= 13 years of age with a CD4+ cell count <= 200 cells/mm3. Patients < 13 years of age with a CD4% <= 14% or a 50% decrease in CD4% in the past 6 months if the previous CD4% was >=20%.
* Patient has failed or is intolerant to currently approved treatments for HIV-1 infection and is unable to participate in a controlled viramune clinical trial.
* Written and informed consent from a parent or guardian for patients < 18 years of age.
* Patient or guardian is willing and able to follow protocol requirements. (PER AMENDMENT 1/29/97:
* Enrollment is closed to adults, as of Jan. 29th only pediatric patients will be enrolled.)

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

Patient qualifies for participation in an actively accruing Viramune controlled clinical trial.

Concurrent Medication:

Excluded:

* Dicumarol, Warfarin, and other anticoagulant medications.
* Tolbutamide.
* Investigational drugs, all protease inhibitors, and all other non-nucleoside transcriptase inhibitors.
* Neurotoxic drugs.
* Cimetidine.
* Erythromycin.

Required:

Patient has failed or is intolerant to currently approved treatments for HIV-1 infection.

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Boehringer Ingelheim Pharmaceuticals Inc, Ridgefield, Connecticut, United States